CLINICAL TRIAL: NCT06313905
Title: DRYLESS: Randomized Controlled Trial of EVADRY® vs Placebo in the Treatment of Xerostomia in Sjögren's Syndrome
Brief Title: EVADRY® in the Treatment of Xerostomia in Sjögren's Syndrome
Acronym: DRYLESS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Fatma Said, Associate professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRYLESS1; CHU La Rabta (Other: La Rabta hospital)
Record Dates: First submitted 2024-03-02; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Sjogren's Syndrome
Keywords: xerostomia; sjogren's syndrom; treatment
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia

STUDY DESIGN:
Intervention Model Description: double-blind randomized study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVADRY (Experimental): 90 Sjogren's syndrom patients with objective xerostomia receiving the EVADRY dietary supplement treatment.
  Interventions: Dietary Supplement: EVADRY
- PLACEBO (Placebo Comparator): 90 Sjogren's syndrom patients with objective xerostomia receiving a placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: EVADRY — The EVADRY oral spray and the placebo are produced by Wellnet laboratory.
  • EVADRY spray: It is a phytotherapy-based medication in the form of an oral spray. It is a 100 ml bottle containing ALEO BARBADENSIS LEAF WATER (1 ml), Chamomilla Recutita Flower extract (30 mg), TOCOPHEROL (10 mg), hyaluronic acid (2 mg), mentha spicata herb oil (10 mg), and eugenol (40 µg).
  Arms: EVADRY
Other: Placebo — The placebo corresponds to flavored water (mint extract) with the same taste as EVADRY. It is placed in a bottle with the same appearance as EVADRY.
  Both products are administered at a rate of 5 intra-oral sprays per day.
  Arms: PLACEBO

SUMMARY:
Xerostomia is a common and very bothersome manifestation that impairs the quality of life in Sjogren's syndrome. Symptomatic therapeutic alternatives for this syndrome are limited in Tunisia. We resort to bromhexine off-label with low efficacy. The aim of this work is to demonstrate the superiority of a treatment based on dietary supplements (EVADRY) vs placebo in the treatment of xerostomia. This is a double-blind randomized clinical trial with 2 arms: an EVADRY arm (n=90) and a placebo arm (n=90). The primary outcome measure is a 35% increase in salivary flow after 3 months. Secondary outcome measures were based on the Oral Health Impact Profile questionnaire, Xerostomia Inventory, the HAD depression scale, and the buccal Schirmer test.

DETAILED DESCRIPTION:
Study design:

This is a randomized controlled double-blind clinical trial involving 2 groups:

* Group 1: consisting of 90 patients receiving the EVADRY dietary supplement treatment.
* Group 2: consisting of 90 patients receiving a placebo

Inclusion and exclusion criteria:

• Inclusion criteria:

The included patients meet the following criteria:

* age over 18 years
* diagnosis of Sjogren's syndrome according to ACR/EULAR 2016 criteria
* continuous xerostomia for more than 3 months
* initial salivary flow rate < 0.1 ml/min

  • Non-inclusion criteria:
* allergy or hypersensitivity to any of the products
* pregnancy
* breastfeeding
* oral or throat surgery before wound healing
* cognitive or dementia disorders

  * Exclusion criteria:

These include:

* Occurrence of cognitive or dementia disorders
* Pregnancy
* Allergy to any of the components of the EVADRY product
* Indication of oral or throat surgery

Randomization:

This is a randomization by random blocks. A co-investigator (who is not in contact with the patients) will be responsible for this randomization. The EVADRY treatment and the placebo will have the same packaging. Codes will be assigned to the sprays by the investigator responsible for the randomization. These codes will be placed in sealed envelopes and will only be opened at the end of the study. They will be kept by another investigator who has no knowledge of the randomization.

Treatment and interventions:

The EVADRY oral spray and the placebo are produced by Wellnet laboratory.

• EVADRY spray: It is a phytotherapy-based medication in the form of an oral spray. It is a 100 ml bottle containing ALEO BARBADENSIS LEAF WATER (1 ml), Chamomilla Recutita Flower extract (30 mg), TOCOPHEROL (10 mg), hyaluronic acid (2 mg), mentha spicata herb oil (10 mg), and eugenol (40 µg).

* The placebo corresponds to flavored water (mint extract) with the same taste as EVADRY. It is placed in a bottle with the same appearance as EVADRY.

Both products are administered at a rate of 5 intra-oral sprays per day.

Evaluation criteria:

• Primary evaluation criterion: It is based on the measurement of salivary flow rate (SFR). It consists of asking the patient to collect their saliva in the morning without prior stimulation (no smoking, chewing gum, or alcohol one hour before) in a graduated tube for 15 minutes. The patient should be comfortably seated with their head slightly tilted forward and their mouth open to allow saliva to flow. A value less than 0.1 ml/minute corresponds to hyposalivation.

• Secondary evaluation criteria:

* Xerostomia Inventory in French version: it is a questionnaire composed of 11 questions. For each item, there is an evaluation of its frequency (never, rarely, occasionally, quite often, very often). The total score ranges from 11 to 55 points.
* OHIP-14 questionnaire: it includes 7 dimensions with 14 items to assess quality of life. The higher the score on this questionnaire, the more negative the impact on quality of life.
* HAD scale: it is an instrument that allows screening for anxiety and depressive disorders. It consists of 14 items rated from 0 to 3 : 7 for anxiety and 7 for depression. We will have 2 scores. A score ≤7 corresponds to the absence of symptoms, ≥11 corresponds to definite symptomatology, and between the two, it is doubtful.
* Buccal Schirmer test: it consists of a strip of Whatman paper (blotting paper) placed in a polyethylene bag, with the first 5 mm of the strip protruding from one end of the bag. This end is then folded and placed under the patient's tongue in contact with the floor of the mouth for 5 minutes. The patient should be in a forward-leaning position, hands on knees, and eyes closed. After five minutes, the strip is removed and the soaked portion is measured in centimeters.

Patient follow-up:

The patients will be interviewed and examined initially. During this consultation, the patient's epidemiological and clinical data will be collected. During the same consultation, SFR and buccal Schirmer test will be measured, and Xerostomia Inventory, OHIP-14, and HAD will be calculated.

These tests will be repeated at 1, 2, and 3 months.

Interruption and end of the trial:

Patient follow-up is planned for 3 months. The statistical study is planned for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* diagnosis of Sjogren's syndrome according to ACR/EULAR 2016 criteria
* continuous xerostomia for more than 3 months
* initial salivary flow rate < 0.1 ml/min

Exclusion Criteria:

* Occurrence of cognitive or dementia disorders
* Pregnancy
* Allergy to any of the components of the EVADRY product
* Indication of oral or throat surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
salivary flow rate (SFR) | at inclusion, after 1, 2 and 3 months
  It consists of asking the patient to collect their saliva in the morning without prior stimulation (no smoking, chewing gum, or alcohol one hour before) in a graduated tube for 15 minutes. The patient should be comfortably seated with their head slightly tilted forward and their mouth open to allow saliva to flow. A value less than 0.1 ml/minute corresponds to hyposalivation.

SECONDARY OUTCOMES:
Xerostomia Inventory in French version | at inclusion, after 1, 2 and 3 months
  it is a questionnaire composed of 11 questions. For each item, there is an evaluation of its frequency (never, rarely, occasionally, quite often, very often). The total score ranges from 11 to 55 points
Oral Health-related quality of life (OHIP-14) questionnaire | at inclusion, after 1, 2 and 3 months
  it includes 7 dimensions with 14 items to assess quality of life. The higher the score on this questionnaire, the more negative the impact on quality of life
Hospital anxiety and depression (HAD) scale | at inclusion, after 1, 2 and 3 months
  it is an instrument that allows screening for anxiety and depressive disorders. It consists of 14 items rated from 0 to 3 : 7 for anxiety and 7 for depression. We will have 2 scores. A score ≤7 corresponds to the absence of symptoms, ≥11 corresponds to definite symptomatology, and between the two, it is doubtful
Buccal Schirmer test | at inclusion, after 1, 2 and 3 months
  it consists of a strip of Whatman paper (blotting paper) placed in a polyethylene bag, with the first 5 mm of the strip protruding from one end of the bag. This end is then folded and placed under the patient's tongue in contact with the floor of the mouth for 5 minutes. The patient should be in a forward-leaning position, hands on knees, and eyes closed. After five minutes, the strip is removed and the soaked portion is measured in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Ines Naceur, Study Chair — Centre Hospitalo-Universitaire La Rabta; Tayssir Ben Achour, Study Chair — Centre Hospitalo-Universitaire La Rabta; Mayssam Jridi, Study Chair — Centre Hospitalo-Universitaire La Rabta; Monia Smiti, Study Director — Centre Hospitalo-Universitaire La Rabta

IPD SHARING:
Plan to Share IPD: No
all investigators work in the same department